CLINICAL TRIAL: NCT01774227
Title: A Randomized Trial of the Pops-titration Versus the Slow-coagulation Energy Delivery Technique on the Outcome of Diode Laser Transcleral Cyclophotocoagulation in Treatment of Neovascular Glaucoma With Dark Iris
Brief Title: the Pops-titration Versus the Slow-coagulation Cyclophotocoagulation in Treatment of Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Dr.Weerawat Kiddee, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 56-094-02-1-2
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Glaucoma; Intraocular Pressure
Keywords: Refractory glaucoma; Transcleral cyclophotocoagulation (TSCPC); Dark iris; Pops-titration; Slow-coagulation; Neovascular glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Neovascular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The pops-titration group (Experimental): The titration method uses power that is titrated according to the audible "pop".
  Interventions: Procedure: The pops-titration group
- The slow-coagulation group (Experimental): The slow-coagulation group utilize the low-energy using the Gaasterland's slow-coagulation technique
  Interventions: Procedure: The slow-coagulation group

INTERVENTIONS:
Procedure: The pops-titration group — The energy delivery is started at a low level and is increased in intervals till an audible pop is heard, following which the power is reduced downward until the pops are no longer audible, then the treatment is completed at these parameters
  Arms: The pops-titration group
Procedure: The slow-coagulation group — The Gaasterland's slow-coagulation energy delivery technique using the lower power for the longer duration.
  Arms: The slow-coagulation group

SUMMARY:
* Transcleral cyclophotocoagulation (TSCPC) has long been used as refractory glaucoma management and is very easy to learn and easy to perform.
* Recent advances in laser technology; the role of TSCPC is being expanded because it has benefits of noninvasive glaucoma procedure.
* The titration (pops), the fixed high-energy, and the fixed-low energy (slow-coagulation) are three energy delivery techniques.
* The present study would report on the outcome (efficacy and safety) of the slow-coagulation versus the titration method in treatment of refractory glaucoma with dark iris.
* The results would provide reliable evidences to supplement clinical judgment when making a decision in favor of each treatment method for glaucoma patients.

DETAILED DESCRIPTION:
* Several protocols afford delivery of the "optimum" dose of laser energy per session necessary to achieve a long-term effective ocular hypotensive response balancing risks related to a high energy treatment and risks related to retreatment due to suboptimum dose delivery.
* There are two main approaches to delivering laser energy, the pops-titration method and the fixed energy method that are the fixed-high and low-energy (the Gaasterland's slow-coagulation technique).
* Of particular interest is which laser energy delivery method (slow-coagulation versus pops-titration) affords the optimal dose of photocoagulation necessary to achieve an effective long-term intraocular pressure (IOP) reduction while minimizing the risk of adverse events related to overtreatment and retreatments especially in refractory glaucomatous eyes with dark iris color.

ELIGIBILITY:
Inclusion Criteria:

* Refractory glaucoma (Neovascular glaucoma) with
* Eyes with no visual potential and very high intraocular pressure (on maximal medical treatment) in which the intraocular pressure will probably cause corneal complications
* Eyes with no visual potential and very high intraocular pressure (on maximal medical treatment) in which the intraocular pressure cause eye pain and need pain relief
* Eyes with minimal useful vision and intraocular pressure over the target intraocular pressure
* Eyes in which trabeculectomy with mitomycin-C and/or drainage implants have a high probability of failure
* Eyes in which trabeculectomy with mitomycin-C and/or drainage implants have previously failed
* Patient refuses to undergo more aggressive intraocular surgery
* Patients whose general medical condition precludes invasive surgery

Exclusion Criteria:

* The visual acuity in the fellow eye is no light perception
* Have previously been treated by the transcleral cyclophotocoagulation
* Allergy to anesthetic medication
* Can not measure the intraocular pressure by the applanation method

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-05; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Success rate | 60 months
  Success rate defined as the proportion of eyes achieving an intraocular pressure between 6 and 21mmHg with or without topical antiglaucoma medication at the final follow up visit.

SECONDARY OUTCOMES:
Response rate | 60 months
  Response rate defined as the proportion of eyes achieving an intraocular pressure between < 22 mmHg or > 30% drop in an intraocular pressure with or without topical antiglaucoma medication at the final follow up visit.
Cyclodiode efficacy index | 60 months
  Cyclodiode efficacy index defined as the ratio of response rate to the mean number of the treatment session.
Failure rate | 60 months
  Failure rate defined as the proportion of eyes developed hypotony or phthisis bulbi or need to repeat treatment for more than 2 laser sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Kiddee, MD, Study Director — Prince of Songkla University
Locations (1):
- Ophthalmology Department, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Kiddee W, Kittigoonpaisan K, Leelaprasasne S, Tanjana A. Randomized clinical trial for pop titrated versus the slow coagulation cyclophotocoagulation in treating dark irises neovascular glaucoma. Sci Rep. 2025 Aug 18;15(1):30238. doi: 10.1038/s41598-025-16306-9. PMID 40826269